CLINICAL TRIAL: NCT06589414
Title: Reintegrating a Systematic Review Consultation With the General Practitioner After the Cancer Diagnosis Has Been Announced Into the Complex Cancer Patient Pathway: Feasibility Study
Acronym: DAMeGe
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24 GENE 07; ID RCB Number: 2024-A00415-42 (Other: ANSM)
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumours
Keywords: Solid Tumours; Announcement system; General practitioner

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DAMeGe protocol (Other)
  Interventions: Other: Patient care according to the DAMeGe protocol (organisation of a summary consultation with the GP)

INTERVENTIONS:
Other: Patient care according to the DAMeGe protocol (organisation of a summary consultation with the GP) — A summary consultation with the patient's general practitioner (GP) will take place within 15 days of the consultation to announce the cancer diagnosis. This patient-general practitioner consultation will complement the initial consultation.
  At the end of the summary consultation, the patient's satisfaction and that of the GP will be assessed using satisfaction questionnaires.
  In addition, patients will be asked to complete a "patient diary" for the duration of their participation in the study (6 months), in order to record the dates of consultations with the GP and the dates of consultations and/or hospitalisations at the referral care centre.

SUMMARY:
This is a prospective, multicentric, regional study designed to assess the feasibility of setting up a summary consultation with a general practitioner (GP) to complement the consultation for the announcement of a cancer diagnosis.

171 patients will be included in the study.

Each patient will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient with a solid tumour whatever the organ.
3. Patient treated in one of the participating centres as part of a system for announcing the diagnosis of a solid cancer.
4. Patient undergoing cancer treatment in one of the participating centres.
5. Patient with a registered general practitioner in the Occitanie region.
6. Patient affiliated to a French Social Security scheme.
7. Patient having signed informed consent prior to inclusion in the study and prior to any specific procedure for the study.

Exclusion Criteria:

1. Patient already included in another clinical trial concerning a care pathway.
2. Patient deprived of liberty or under legal protection (curatorship and guardianship, safeguard of justice).
3. Pregnant or breast-feeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The ratio between the number of patients who attended the summary consultation with the general practitioner within 15 days of being diagnosed with cancer in the referral care centre and the total number of patients included in the study. | 21 months after the start of the study

SECONDARY OUTCOMES:
The reasons why the summary consultation with the GP did not take place within 15 days of the consultation to announce the cancer diagnosis. | 21 months after the start of the study
  It will be assessed for each patient included in the study in conjunction with the patients or GPs: patient refusal, GP refusal, cancelled or postponed by the patient, cancelled or postponed by the GP, out of time (>15 days), other reason.
The type of consultations carried out with the GP (physical consultations, teleconsultations or home visits) will be presented as follows, using standard descriptive statistics. | 21 months after the start of the study
The number of cancellations of consultations with GPs will be presented as follows, using standard descriptive statistics. | 21 months after the start of the study
The number of postponed consultations with the GP will be presented as follows, using standard descriptive statistics. | 21 months after the start of the study
The overall compliance will be presented as follows, using standard descriptive statistics. | 21 months after the start of the study
The participation will be assessed. | 18 months after the start of the study
  All ratios complementary to the main criterion will be collected and analysed (the number of patients who received the offer to participate in the systematic consultation, the number of patients actually included).
The socio-demographic characteristics of the patients included will be described and analysed. | 21 months after the start of the study
The rate of patients with a change in management between the treatment proposed at the RCP (Multidisciplinary Consultation Meeting) and that carried out in the centre. | 6 months for each patient
  It will be presented in the following format: number, percentage and 95% confidence interval (exact binomial distribution).
The number of hospital admissions and unscheduled consultations at the referral centre during the 6 months of follow-up will be assessed for each patient included in the study. | 6 months for each patient
The satisfaction of patients included in the study and of GPs whose patients take part in the study. | 21 months after the start of the study
  It will be assessed using questionnaires. Responses to the questions will be based on a Likert scale of 1 to 4: 'Completely satisfactory', 'Somewhat satisfactory', 'Somewhat unsatisfactory', 'Not at all satisfactory'.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CH Auch, Auch
  - CH Carcassonne, Carcassonne
  - CHU Larrey, Toulouse
  - CHU Rangueil, Toulouse
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse